CLINICAL TRIAL: NCT05201079
Title: A Randomised, Controlled, Open-label Phase III Clinical Trial in Patients With Primary or Recurrent Clostridioides Difficile (CD) Infection, to Evaluate the Efficacy and Safety of Capsules of Lyophilised Faecal Microbiota vs Fidaxomicin.
Brief Title: Primary or Recurrent Clostridioides Difficile Infection Treatment With Capsules of Lyophilised Faecal Microbiota vs Fidaxomicin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mikrobiomik Healthcare Company S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICD-01; 2020-004591-17 (EudraCT Number)
Record Dates: First submitted 2021-12-14; First posted 2022-01-21 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Clostridium Difficile Infection; Primary Clostridium Difficile Infection
Keywords: Clostridium difficile; FMT; Fecal Microbiota Transfer
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation; Fidaxomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBK-01 (Experimental): Participants will receive MBK-01 capsules of fecal microbiota coming from healthy donors (45 patients).
  Interventions: Biological: MBK-01
- Fidaxomicin (Active Comparator): Participants will receive Fidaxomicin (47 patients).
  Interventions: Drug: Fidaxomicin

INTERVENTIONS:
Biological: MBK-01 — A single dose of 4 capsules of MBK-01 (heterologous lyophilized fecal microbiota coming from healthy donors) orally.
  Other Names: Fecal microbiota transfer
  Arms: MBK-01
Drug: Fidaxomicin — Oral administration of 200mg/12 hours of fidaxomicin for 10 days.
  Other Names: Dificlir; Dificid
  Arms: Fidaxomicin

SUMMARY:
Patients with microbiota alterations developed after being exposed to antibiotics are especially susceptible to Clostridioides difficile infections (CDI). The incidence and severity of CDI has increased in recent years and CDI recurrences (r-CDI) due to the appearance of new episodes in patients with a previous cured CDI, represent a serious and complex clinical issue. Although antibiotics are the recommended therapy for the first episode of CDI, treatment with oral vancomycin and/or metronidazole often results in significant treatment failure. In addition, the treatment of r-CDI is not adequately standardized, and although the most widely used treatment is the administration of fidaxomicin and bezlotoxumab, its efficacy in patients who already have r-CDI is not proven. In the late years, Fecal Microbiota Transfer (FMT) has emerged as the preferred non-pharmacological treatment to manage CDI with multiple recurrences and recent clinical trials have evaluated its potential efficacy and safety in the treatment of patients with primary CD infection.

The objective of this study is to assess the efficacy and safety of the MBK-01 medication, consisting of heterologous lyophilized fecal microbiota capsules coming from healthy donors in comparison to the treatment with fidaxomicin, in 92 patients with primary or r-CDI.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, controlled and open label clinical trial in which patients who suffered an episode of Clostridioides difficile infection (either the first episode or subsequent recurrences) will be randomly assigned (1:1) to one of the following arms:

* Fidaxomicin
* MBK-01 (heterologous lyophilized fecal microbiota)

Objective: To assess the efficacy of FMT with capsules of lyophilized fecal microbiota (MBK-01), compared to the control (fidaxomicin) at 8 weeks after the start of the treatment. Also, assess the safety of MBK-01 and the quality of life of patients participating in the study.

Follow up: participants will return for clinic visits at 72 hours, week 3 and week 8 after the start of the treatment, and will receive follow-up phone calls at month 3 and month 6 after the start of the treatment. Stool samples will be collected from participants for further studies at time 0 and week 8 after the start of the treatment. Study Outcomes are detailed in the specific section of this website.

Rationale: The transferred microbiota restores the recipient's intestinal microbiota by reintroducing bacterial taxa that were absent or in low proportion in the recipient before the FMT. This supports the expansion of the recipient's own commensal microbiota and re-establishing a microbiota community with a high biodiversity.

Donors: All donors are screened to ensure they meet the strict requirements necessary to maintain the safety of the MBK-01.

Justification: The treatment of Clostridioides difficile infections (CDI) with antibiotics is usually effective for acute symptoms, but after the initial treatment, the probability of recurrence at 8 weeks ranges from 10-20 % of cases, and once a patient has a recurrence, the probability of further recurrences increases up to 40-65 %. In recent years, Fecal Microbiota Transfer (FMT) has emerged as the preferred non-pharmacological treatment to manage CDI with multiple recurrences and recent clinical trials have evaluated its potential efficacy and safety in the treatment of patients with primary CD infection. Although antibiotics are the recommended therapy for the first episode of CDI, treatment with oral vancomycin and/or metronidazole often results in significant treatment failure, with recurrences occurring in up to 30-40% of patients. Furthermore, antibiotic treatment does not correct deficiencies in the intestinal microbiota that facilitate CD infection and is associated with the risk of the emergence of antibiotic-resistant bacteria. Moreover, the treatment of recurrences is not adequately standardized. In recent years, although the most widely used alternatives have been fidaxomicin and bezlotoxumab, their efficacy in patients who already suffer from r-CDI is not proven. The administration of the FMT through oral capsules, although it is not standardized, has proven to be effective in the restoration of intestinal microbiota of patients with r-CDI. In addition, the use of lyophilized formulas facilitates the concentration of bacteria and further optimizes the donors' sample and reduces the amount of capsules that the patient has to ingest.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders, over 18 years.
2. Patients that undergo an episode of CD infection (either the first episode or subsequent recurrences).
3. Presence of an episode of diarrhea defined as ≥3 stools/24 hours, at the beginning of the episode.
4. Confirmation of the presence of CD toxin A and/or B in faeces, by a direct toxin detection test or by the PCR technique for the detection of toxin/s producing genes, at the start of the episode that is going to be treated in the clinical trial (the toxin test must be positive within 7 days prior to the enrolment of the patient in the trial).

Exclusion Criteria:

1. Previous faecal microbiota transfer.
2. Transplanted patients, except those with a solid organ transplant of more than 2 years, with good organ function.
3. Absolute neutrophil count <500 cells /μL at the time of the enrollment in the study.
4. Pregnancy, breastfeeding, or pregnancy intentions over the course of the study.
5. Active treatment with bile acid sequestrants (for instance: cholestyramine).
6. Positive patients for the human immunodeficiency virus (HIV) except those with lymphocytes T CD4 count > 200 cells/μL and viral load less than 20 copies.
7. Swallowing dysfunction or no oral motor coordination.
8. Patient admitted in an intensive care unit or expected to be admitted in an intensive care unit due to serious illness.
9. History of significant medical conditions that, in the opinion of the investigator, would not allow an adequate evaluation or follow-up of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cobo, MD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (21):
- Spain (21):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Quirónsalud Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Josep Trueta de Gerona, Girona
  - Hospital San Pedro, Logroño
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Universitario de Araba, Vitoria-Gasteiz
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Reigadas E, Bouza E, Olmedo M, Vazquez-Cuesta S, Villar-Gomara L, Alcala L, Marin M, Rodriguez-Fernandez S, Valerio M, Munoz P. Faecal microbiota transplantation for recurrent Clostridioides difficile infection: experience with lyophilized oral capsules. J Hosp Infect. 2020 Jun;105(2):319-324. doi: 10.1016/j.jhin.2019.12.022. Epub 2019 Dec 26. PMID 31883938
- [Background] Reigadas E, Olmedo M, Valerio M, Vazquez-Cuesta S, Alcala L, Marin M, Munoz P, Bouza E. Fecal microbiota transplantation for recurrent Clostridium difficile infection: Experience, protocol, and results. Rev Esp Quimioter. 2018 Oct;31(5):411-418. Epub 2018 Sep 14. PMID 30221898
- See also: EU Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2020-004591-17/ES

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was recruited on 29th October 2021. Last patient was recruited on 15th November 2023. Patients were recruited in the study sites.
Pre-assignment Details: One selected patient was excluded before randomisation because of screening failure.
Groups:
- Fidaxomicin: Participants will receive Fidaxomicin (47 patients). Dificlir: Oral administration of 200mg/12 hours of fidaxomicin for 10 days.
Period: Overall Study
Arm/Group | MBK-01 | Fidaxomicin
Started | 45 | 47
Completed | 23 | 25
Not Completed | 22 | 22
Not completed — Adverse Event | 7 | 11
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Forbidden medication | 9 | 5
Not completed — Transfer to another hospital | 0 | 1
Not completed — Clinical condition | 1 | 0
Not completed — SAE and sepsis | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention To Treat (ITT) population: all patients randomized in the study, whether or not they fulfil inclusion/exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | MBK-01 | Fidaxomicin | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.22 (17.24) | 65.26 (14.65) | 65.24 (15.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 15 | 17 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 44 | 45 | 89
  Amerindian | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Spain | 45 | 47 | 92
Medical history: number of previous pathologies [Mean (Standard Deviation); unit: previous pathologies] | 7.96 (4.79) | 6.62 (4.33) | 7.27 (4.58)
Medical history: number of pretreatments [Mean (Standard Deviation); unit: pretreatments] | 2.33 (2.00) | 2.51 (2.34) | 2.38 (2.30)
Clostridioides difficile infection episode [Count of Participants; unit: Participants]
  Primary episode | 25 | 28 | 53
  Recurrent episode | 20 | 19 | 39
Previous antibiotic treatment [Count of Participants; unit: Participants] — A pre-washing out period before the administration of the study treatment was mandatory for all patients who received previous antibiotic Population: In patients who received previous antibiotic treatment, the number of patients that carried out a pre-washing out period was analyzed.
  Participants
    Previous antibiotic: Yes | 23 | 29 | 52
    Previous antibiotic: No | 22 | 18 | 40
    Pre-washing out: number analyzed (Participants) | 23 | 29 | 52
    Pre-washing out: Yes | 23 | 29 | 52
    Pre-washing out: No | 0 | 0 | 0
Duration of antibiotic treatment [Mean (Standard Deviation); unit: days] — Population: n patients who received previous antibiotic treatment, the duration of the antibiotic treatment was analyzed.
  days
    number analyzed (Participants) | 23 | 29 | 52
    (all) | 2.96 (1.72) | 3.21 (1.15) | 3.08 (1.41)
Proton pump inhibitor treatment [Count of Participants; unit: Participants]
  Yes | 26 | 28 | 54
  No | 19 | 19 | 38
SF36 Questionnaire (The Short Form-36 Health Survey) to Evaluate the Quality of Life [Mean (Standard Deviation); unit: units on a scale] — For each dimension (physical functioning, role limits-physical, bodily pain, general health, vitality, social functioning, role limits-emotional, mental health), the scale ranges from 0 (the worst health status for that dimension) to 100 (the best health status). Population: SF36 Questionnaire analysis was conducted in the population that completed the questionnaire
  units on a scale
    Physical function: number analyzed (Participants) | 41 | 46 | 87
    Physical function | 56.90 (35.90) | 57.07 (33.71) | 56.99 (34.57)
    Physical role: number analyzed (Participants) | 41 | 46 | 87
    Physical role | 33.48 (33.44) | 36.55 (32.81) | 35.90 (32.96)
    Bodily pain: number analyzed (Participants) | 41 | 46 | 87
    Bodily pain | 52.91 (29.84) | 57.25 (29.07) | 55.18 (29.35)
    General health: number analyzed (Participants) | 41 | 46 | 87
    General health | 55.13 (17.07) | 54.85 (20.62) | 54.98 (18.90)
    Vitality: number analyzed (Participants) | 41 | 46 | 87
    Vitality | 38.33 (11.75) | 35.69 (18.56) | 37.02 (15.74)
    Social function: number analyzed (Participants) | 41 | 46 | 87
    Social function | 65.08 (15.53) | 63.77 (19.02) | 64.39 (17.36)
    Emotional role: number analyzed (Participants) | 41 | 46 | 87
    Emotional role | 58.13 (38.98) | 68.30 (32.18) | 63.51 (35.70)
    Mental health: number analyzed (Participants) | 41 | 46 | 87
    Mental health | 54.64 (16.93) | 56.06 (17.17) | 55.40 (16.97)
Declared outcome of health [Mean (Standard Deviation); unit: units on a scale] — Declared outcome of health measured by SF36 questionnaire. The declared outcome of health is a transition item in The Short Form-36 Health Survey (SF-36). The results are measured as follows: 1 (excellent), (2) very good, 3 (good), 4 (regular) and 5 (poor). Population: Outcome analysis was conducted on the population that completed the SF36 questionnaire
  units on a scale
    number analyzed (Participants) | 42 | 46 | 88
    (all) | 3.74 (1.01) | 3.65 (0.97) | 3.69 (0.99)

OUTCOME MEASURES:

1. Primary Outcome: Global Absence of Diarrhea Due to Clostridiodes Difficile 8 Weeks After the Start of the Treatment
Description: Number of patients who showed recurrence of at least one Episode of Diarrhea (3 or More Stools/24 Hours) 8 Weeks After the Start of the Treatment. Recurrence is understood as the reappearance of clinical manifestations of a new episode of CDI that re-occurs within 8 weeks after the onset of symptoms of a previous episode that was resolved.
Time Frame: 8 weeks after the start of the treatment
Population: For the analysis of recurrences, there are 77 patients evaluable. The remaining patients were excluded from this analysis due to different reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 37 | 40
Participants | 4 | 9
Statistical Analysis 1: Comparison: MBK-01 vs Fidaxomicin; Test type: Superiority; p = 0.228, Regression, Logistic — Alpha: 0.0221; Odds Ratio (OR) = 2.395, 97.79% CI 2-sided [0.540 to 10.624] — Numerator: fidaxomicin; denominator: MBK-01

2. Primary Outcome: Absence of Diarrhea: Number of Episodes of Diarrhea (3 or More Stools/24 Hours) 72 Hours After the Start of the Treatment
Description: Diarrhea resolution: <3 stools/24 hours for at least 2 consecutive days after the end of the treatment.
Time Frame: 72 hours after the start of the treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 37 | 40
Participants | 1 | 0

3. Primary Outcome: Absence of Diarrhea: Number of Episodes of Diarrhea (3 or More Stools/24 Hours) 3 Weeks After the Start of the Treatment
Description: Diarrhea resolution: <3 stools/24 hours for at least 2 consecutive days after the end of the treatment.
Time Frame: 3 weeks after the start of the treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 37 | 40
Participants | 2 | 2

4. Primary Outcome: Absence of Diarrhea: Number of Episodes of Diarrhea (3 or More Stools/24 Hours) 3 Months After the Start of the Treatment
Description: Diarrhea resolution: <3 stools/24 hours for at least 2 consecutive days after the end of the treatment.
Time Frame: 3 months after the start of the treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 37 | 40
Participants | 4 | 9

5. Primary Outcome: Absence of Diarrhea: Number of Episodes of Diarrhea (3 or More Stools/24 Hours) 6 Months After the Start of the Treatment
Description: Diarrhea resolution: <3 stools/24 hours for at least 2 consecutive days after the end of the treatment.
Time Frame: 6 months after the start of the treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 37 | 40
Participants | 4 | 9

6. Secondary Outcome: Duration of Hospitalisation
Description: Time, in days, that the patient remains in the hospital as a result of CDI (but not necessarily indicating a recurrence of diarrhea due to CDI).
Time Frame: Up to 8 weeks after the start of the treatment
Population: Out of all partipants analyzed, only 14 in the MBK-01 group and 6 in the fidaxomicin group where hospitalised due to CDI. No participant received both treatments in any case.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
days | 6.50 [4.00 to 8.00] | 5.50 [5.00 to 6.75]

7. Secondary Outcome: Good/Bad Progress of the Patient
Description: A bad progress of the patient is defined as the detection 48-72 hours after the start of the treatment (MBK-01 or Fidaxomicin) of:
  A worsening of the diarrhea episode (at least one stool more than at baseline, baseline being understood as the time of the start of the study treatment (fidaxomicin or MBK01)).
  And, at least, one of the following factors:
  * Increase in C-reactive protein (CRP) value (> 5 % of the baseline value).
  * Increase in white blood cell count (> 5 % of the baseline value).
  * Progression to sepsis: hypotension or organ failure with no other apparent cause.
Time Frame: Up to 72 hours after the start of the treatment
Population: The analysis is carried out on ITT population, excluding patients with no data related to this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 43 | 45
Participants
  Good progress | 43 | 44
  Bad progress | 0 | 1
  Worsening of the diarrhea episode | 2 | 1
  Increase in CRP value: number analyzed (Participants) | 40 | 42
  Increase in CRP value | 3 | 3
  Increase in white blood cell count: number analyzed (Participants) | 39 | 36
  Increase in white blood cell count | 7 | 8
  Progression to sepsis | 0 | 0
Statistical Analysis 1: Comparison: MBK-01 vs Fidaxomicin; Alpha value used: 0.0221; Test type: Superiority; Statistical analysis using Odds Ratio cannot be performed because there are zero patients with bad progress in MBK-01 group

8. Secondary Outcome: Time to Recurrence Depending on Randomisation Groups
Description: Recurrence: Reappearance of clinical manifestations of a new CDI episode in a patient with an CDI episode treated and cured in the previous 8 weeks.
Time Frame: Up to 6 months after the start of the treatment
Population: For the analysis of time to recurrence, there were 77 evaluable participants (37 in MBK-01 and 40 in fidaxomicin group). The reasons for non-evaluable were:
  MBK-01:
  * Non-evaluable (n=8)
  * Death (n=1)
  * Forbidden medication (n=2)
  * Investigator decision (n=1)
  * Adverse event (n=3)
  * Informed consent withdrawal (n=1)
  Fidaxomicin:
  * Non-evaluable (n=7):
  * Death (n=1)
  * Forbidden medication (n=2)
  * Investigator decision (n=1)
  * Adverse event (n=2)
  * Transfer to other hospital (n=1)
Measure: Mean (Standard Error); unit: weeks
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 37 | 40
weeks | 24.70 (1.34) | 22.40 (1.53)
Statistical Analysis 1: Comparison: MBK-01 vs Fidaxomicin; Test type: Superiority; p = 0.300, Regression, Cox — Alpha: 0.0221; Degrees of freedom: 1; Score (logrank) test = 1.25

9. Secondary Outcome: Duration of Treatment
Description: Duration in days of the treatment.
Time Frame: Up to 10 days
Population: There are 46 evaluable patients in the Fidaxomicin group because 1 patient assigned to fidaxomicin was transferred to another hospital before first administration of the treatment. No patient received both treatments under any circumstances.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 46
days | 1.0 [1.0 to 1.0] | 10.0 [10.0 to 10.0]

10. Secondary Outcome: Overall Survival
Description: Percentage of patients that are still alive after a defined period of time from the beginning of the treatment.
Time Frame: Up to 6 months after the start of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Participants | 44 | 46
Statistical Analysis 1: Comparison: MBK-01 vs Fidaxomicin; Test type: Superiority; p = 0.900, Regression, Cox — Alpha: 0.0221; Degrees of freedom: 1; Score (logrank) test = 0.02

11. Secondary Outcome: Number of Adverse Events Per Randomisation Group
Description: Number of Adverse Events per randomisation group since baseline.
Time Frame: Up to 6 months after the start of the treatment
Measure: Number; unit: Number of Adverse Events
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Number of Adverse Events | 89 | 103

12. Secondary Outcome: Type of Adverse Events Per Ramdomisation Group
Description: Type of Adverse Events per ramdomisation group since baseline.
Time Frame: Up to 6 months after the start of the treatment
Measure: Number; unit: Number of Adverse Events
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Number of Adverse Events
  Blood and lymphatic system disorders: anaemia | 1 | 0
  Blood and lymphatic system disorders: iron deficiency anaemia | 0 | 1
  Blood and lymphatic system disorders: leukocytosis | 1 | 0
  Cardiac disorders: cardiac failure | 0 | 1
  Ear and labyrinth disorders: vertigo | 1 | 0
  Gastrointestinal disorders: abdominal discomfort | 1 | 2
  Gastrointestinal disorders: abdominal pain | 4 | 3
  Gastrointestinal disorders: abdominal pain lower | 0 | 1
  Gastrointestinal disorders: abdominal pain upper | 1 | 1
  Gastrointestinal disorders: colitis ulcerative | 1 | 0
  Gastrointestinal disorders: constipation | 1 | 2
  Gastrointestinal disorders: dental discomfort | 1 | 0
  Gastrointestinal disorders: diarrhea | 17 | 27
  Gastrointestinal disorders: erosive duodenitis | 0 | 1
  Gastrointestinal disorders: flatulence | 2 | 4
  Gastrointestinal disorders: gastrointestinal sounds abnormal | 0 | 1
  Gastrointestinal disorders: gastrooesophageal reflux disease | 0 | 1
  Gastrointestinal disorders: haemorroids | 2 | 1
  Gastrointestinal disorders: irritable bowel syndrome | 0 | 1
  Gastrointestinal disorders: nausea | 3 | 3
  Gastrointestinal disorders: odynophagia | 1 | 0
  Gastrointestinal disorders: reflux gastritis | 1 | 0
  Gastrointestinal disorders: vomiting | 4 | 2
  General disorders and administration site conditions: fatigue | 0 | 1
  General disorders and administration site conditions: medical device site reaction | 0 | 1
  General disorders and administration site conditions: pain | 3 | 1
  General disorders and administration site conditions: polyp | 0 | 1
  General disorders and administration site conditions: pyrexia | 3 | 2
  Infections and infestations: Clostridium difficile colitis | 0 | 1
  Infections and infestations: Clostridium difficile infection | 2 | 3
  Infections and infestations: COVID-19 | 1 | 1
  Infections and infestations: cystitis | 1 | 1
  Infections and infestations: Escherichia urinary tract infection | 0 | 1
  Infections and infestations: gastroenteritis | 3 | 0
  Infections and infestations: influenza | 1 | 0
  Infections and infestations: oral candidiasis | 1 | 0
  Infections and infestations: perineal abscess | 1 | 0
  Infections and infestations: pneumonia | 0 | 1
  Infections and infestations: respiratory tract infection | 0 | 1
  Infections and infestations: urinary tract infection | 3 | 2
  Injury, poisoning and procedural complications: fall | 1 | 0
  Injury, poisoning and procedural complications: spinal fracture | 0 | 1
  Injury, poisoning and procedural complications: synovial rupture | 1 | 0
  Investigations: blood creatinine increased | 0 | 1
  Investigations: cardiac murmur | 1 | 0
  Investigations: Clostridium test positive | 1 | 0
  Investigations: C-reactive protein increased | 13 | 7
  Investigations: international normalised ratio increased | 0 | 1
  Investigations: white blood cell count increased | 0 | 2
  Metabolism and nutrition disorders: folate deficiency | 0 | 1
  Metabolism and nutrition disorders: hypokalaemia | 0 | 1
  Metabolism and nutrition disorders: hyponatraemia | 0 | 1
  Metabolism and nutrition disorders: vitamin B12 deficiency | 0 | 1
  Metabolism and nutrition disorders: vitamin D deficiency | 0 | 1
  Musculoskeletal and connective tissue disorders: back pain | 1 | 1
  Musculoskeletal and connective tissue disorders: musculoskeletal chest pain | 0 | 1
  Nervous system disorders: dizziness | 0 | 1
  Nervous system disorders: headache | 3 | 4
  Nervous system disorders: migraine | 1 | 0
  Psychiatric disorders: agitation | 1 | 0
  Psychiatric disorders: insomnia | 0 | 1
  Psychiatric disorders: mixed anxiety and depressive disorder | 0 | 1
  Renal and urinary disorders: microalbuminuria | 0 | 1
  Renal and urinary disorders: oliguria | 1 | 0
  Reproductive system and breast disorders: prostatitis | 1 | 0
  Respiratory, thoracic and mediastinal disorders: catarrh | 1 | 0
  Skin and subcutaneous tissue disorders: angioedema | 0 | 1
  Skin and subcutaneous tissue disorders: hidradenitis | 0 | 1
  Skin and subcutaneous tissue disorders: pruritus | 0 | 1
  Skin and subcutaneous tissue disorders: toxic skin eruption | 0 | 1
  Skin and subcutaneous tissue disorders: vascular purpura | 0 | 1
  Surgical and medical procedures: prophylaxis | 1 | 0
  Surgical and medical procedures: tooth extraction | 0 | 1
  Vascular disorders: hot flush | 0 | 1
  Vascular disorders: hypertensive crisis | 1 | 0

13. Secondary Outcome: Number of Serious Adverse Events Per Ramdomisation Group
Description: Number of Serious Adverse Events per ramdomisation group since baseline.
Time Frame: Up to 6 months after the start of the treatment
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Number of Serious Adverse Events | 11 | 5

14. Secondary Outcome: Type of Serious Adverse Events Per Ramdomisation Group
Description: Type of Serious Adverse Events per ramdomisation group since baseline.
Time Frame: Up to 6 months after the start of the treatment
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Number of Serious Adverse Events
  Cardiac disorders: cardiac failure | 1 | 0
  Gastrointestinal disorders: colitis ulcerative | 1 | 0
  Gastrointestinal disorders: diarrhea | 0 | 1
  Gastrointestinal disorders: inflammatory bowel disease | 0 | 1
  Gastrointestinal disorders: intra-abdominal fluid collection | 1 | 0
  Gastrointestinal disorders: rectal haemorrhage | 0 | 1
  Infections and infestations: anal abscess | 1 | 0
  Infections and infestations: Clostridium difficile infection | 1 | 1
  Infections and infestations: necrotising fasciitis | 1 | 0
  Infections and infestations: pneumonia | 1 | 0
  Infections and infestations: pyelonephritis acute | 1 | 0
  Infections and infestations: sepsis | 1 | 0
  Neoplasms, benign, malignant and unspecified (incl cysts and polyps): renal cancer | 1 | 0
  Respiratory, thoracic and mediastinal disorders: acute respiratory distress syndrome | 0 | 1
  Respiratory, thoracic and mediastinal disorders: acute respiratory failure | 1 | 0

15. Secondary Outcome: Adverse Events Related to the Treatment
Description: Adverse Events related to the treatment since baseline.
Time Frame: Up to 6 months after the start of the treatment
Measure: Number; unit: Number of Adverse Events
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Number of Adverse Events | 1 | 3

16. Secondary Outcome: Adverse Event Seriousness
Description: Adverse Event Seriousness since baseline.
Time Frame: Up to 6 months after the start of the treatment
Measure: Number; unit: Number of Adverse Events
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Number of Adverse Events
  Mild | 70 | 77
  Moderate | 17 | 22
  Severe | 1 | 4
  Life threatening | 0 | 0
  Death | 1 | 0

17. Secondary Outcome: Adverse Events Related to the CDI
Description: Adverse Events related to the CDI since baseline.
Time Frame: Up to 6 months after the start of the treatment
Measure: Number; unit: Number of Adverse Events
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Number of Adverse Events
  Clostridium difficile colitis | 0 | 1
  Diarrhea | 17 | 28
  Clostridium difficile infection | 3 | 4
  Positive Clostridium test | 1 | 0
  Total of Adverse Events related to the CDI | 21 | 33

18. Secondary Outcome: Mortality Associated With CDI
Description: Percentage of patients that die due to CDI after a defined period of time from the beginning of the treatment.
Time Frame: Up to 6 months after the start of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Participants | 0 | 0

19. Secondary Outcome: Intensive Care Unit Admissions (ICU)
Description: Percentage of patients admitted in the ICU after a defined period of time from the beginning of the treatment.
Time Frame: Up to 6 months after the start of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Participants | 0 | 0

20. Secondary Outcome: Adverse Events of Special Interest
Description: Adverse Events of special interest since baseline.
Time Frame: Up to 6 months after the start of the treatment
Measure: Number; unit: Number of AEs
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 45 | 47
Number of AEs
  Vomiting | 4 | 2
  Urinary tract infection | 1 | 0
  Pyrexia | 3 | 2
  Prostatitis | 1 | 0
  Perineal abscess | 1 | 0
  Pain | 3 | 1
  Nausea | 3 | 3
  Migraine | 1 | 0
  Irritable bowel syndrome | 0 | 1
  Influenza | 1 | 0
  Inflammatory bowel disease | 0 | 1
  Headache | 2 | 3
  Haemorrhoids | 1 | 0
  Gastroenteritis | 1 | 0
  Flatulence | 1 | 3
  Fatigue | 0 | 1
  Diarrhoea | 17 | 26
  Cystitis | 0 | 1
  Constipation | 1 | 2
  Colitis ulcerative | 1 | 0
  Clostridium test positive | 1 | 0
  Clostridium difficile infection | 3 | 4
  Clostridium difficile colitis | 0 | 1
  COVID-19 | 0 | 1
  C-reactive protein increased | 13 | 5
  Abdominal pain upper | 1 | 1
  Abdominal pain | 4 | 3
  Abdominal discomfort | 0 | 2

21. Secondary Outcome: SF36 Questionnaire (The Short Form-36 Health Survey) to Evaluate the Quality of Life
Description: For each dimension (physical functioning, role limits-physical, bodily pain, general health, vitality, social functioning, role limits-emotional, mental health), the scale ranges from 0 (the worst health status for that dimension) to 100 (the best health status).
Time Frame: Day 0, 8 weeks and 6 months after the start of the treatment
Population: In addition to the lack of some data by different reasons through the study (i.e. dropout due to the use of forbidden medication), not all the patients completed all the visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBK-01 | Fidaxomicin
Number analyzed (Participants) | 42 | 46
score on a scale
  Physical Function (day 0) | 56.9 (35.9) | 57.07 (33.71)
  Physical Function (8 weeks): number analyzed (Participants) | 30 | 31
  Physical Function (8 weeks) | 68.5 (30.6) | 62.58 (30.44)
  Physical Function (6 months): number analyzed (Participants) | 12 | 11
  Physical Function (6 months) | 77.5 (27.01) | 77.73 (27.14)
  Bodily pain (day 0) | 52.91 (29.84) | 57.25 (29.07)
  Bodily pain (8 weeks): number analyzed (Participants) | 30 | 31
  Bodily pain (8 weeks) | 35.19 (29.19) | 40.5 (28.33)
  Bodily pain (6 months): number analyzed (Participants) | 12 | 11
  Bodily pain (6 months) | 35.19 (33.78) | 27.27 (28.27)
  General health (day 0) | 55.13 (17.07) | 54.85 (20.62)
  General health (8 weeks): number analyzed (Participants) | 30 | 31
  General health (8 weeks) | 47.18 (18.04) | 49.13 (17.5)
  General health (6 months): number analyzed (Participants) | 12 | 11
  General health (6 months) | 41.03 (15.5) | 38.46 (16.14)
  Vitality (day 0) | 38.1 (11.52) | 35.69 (18.56)
  Vitality (8 weeks): number analyzed (Participants) | 30 | 31
  Vitality (8 weeks) | 36.39 (17.02) | 40.86 (11.85)
  Vitality (6 months): number analyzed (Participants) | 12 | 11
  Vitality (6 months) | 35.42 (7.22) | 36.36 (8.56)
  Social role (day 0) | 65.08 (15.53) | 63.77 (19.02)
  Social role (8 weeks): number analyzed (Participants) | 30 | 31
  Social role (8 weeks) | 63.33 (14.78) | 63.44 (11.72)
  Social role (6 months): number analyzed (Participants) | 12 | 11
  Social role (6 months) | 59.72 (11.14) | 69.7 (10.05)
  Emotional role (day 0) | 59.13 (39.04) | 68.3 (32.18)
  Emotional role (8 weeks): number analyzed (Participants) | 30 | 31
  Emotional role (8 weeks) | 82.78 (25.7) | 70.43 (28.04)
  Emotional role (6 months): number analyzed (Participants) | 12 | 11
  Emotional role (6 months) | 86.11 (22.29) | 84.09 (20.57)
  Mental health (day 0) | 55.27 (16.92) | 56.06 (17.17)
  Mental health (8 weeks): number analyzed (Participants) | 30 | 31
  Mental health (8 weeks) | 60 (16.42) | 57.83 (13.84)
  Mental health (6 months): number analyzed (Participants) | 12 | 11
  Mental health (6 months) | 63.69 (11.97) | 62.34 (12.81)
  Physical Role (day 0) | 33.48 (33.44) | 36.55 (32.81)
  Physical Role (8 weeks): number analyzed (Participants) | 30 | 31
  Physical Role (8 weeks) | 69.17 (35.84) | 57.46 (30.64)
  Physical Role (6 months): number analyzed (Participants) | 12 | 11
  Physical Role (6 months) | 72.92 (29.95) | 74.43 (34.51)
Statistical Analysis 1: Comparison: MBK-01 vs Fidaxomicin; For each area of the SF-36 questionnaire, a mixed ANOVA for the effect of Group, Visit, and interaction effect of Group x Visit was performed. alpha = 0.0221; Test type: Superiority; p = 0.749, ANOVA — Main effect of the Group for the Physical Function area of the SF-36 questionnaire. F statistic (1,56) = 0.104
Statistical Analysis 2: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.620, ANOVA — Main effect of the Visit for the Physical Function area of the SF-36 questionnaire. F statistic (1,56) = 0.249
Statistical Analysis 3: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.160, ANOVA — Main effect of the Group x Visit interaction for the Physical Function area of the SF-36 questionnaire. F statistic (1,56) = 2.024
Statistical Analysis 4: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.614, ANOVA — Main effect of the Group for the Bodily pain area of the SF-36 questionnaire. F statistic (1,56) = 0.257
Statistical Analysis 5: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.007, ANOVA — Main effect of the Visit for the Bodily pain area of the SF-36 questionnaire. F statistic (1,56) = 7.705. Effect size = 0.046
Statistical Analysis 6: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.718, ANOVA — Main effect of the Group x Visit interaction for the Bodily pain area of the SF-36 questionnaire. F statistic (1,56) = 0.132
Statistical Analysis 7: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.494, ANOVA — Main effect of the Group for the General Health area of the SF-36 questionnaire. F statistic (1,56) = 0.474
Statistical Analysis 8: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.339, ANOVA — Main effect of the Visit for the General Health area of the SF-36 questionnaire. F statistic (1,56) = 0.932
Statistical Analysis 9: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.380, ANOVA — Main effect of the Group x Visit interaction for the General health area of the SF-36 questionnaire. F statistic (1,56) = 0.783
Statistical Analysis 10: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.790, ANOVA — Main effect of the Group for the Vitality area of the SF-36 questionnaire. F statistic (1,56) = 0.072
Statistical Analysis 11: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.498, ANOVA — Main effect of the Visit for the Vitality area of the SF-36 questionnaire. F statistic (1,56) = 0.465
Statistical Analysis 12: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.023, ANOVA — Main effect of the Group x Visit interaction for the Vitality area of the SF-36 questionnaire. F statistic (1,56) = 5.490
Statistical Analysis 13: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.553, ANOVA — Main effect of the Group for the Social role area of the SF-36 questionnaire. F statistic (1,56) = 0.356
Statistical Analysis 14: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.718, ANOVA — Main effect of the Visit for the Social role area of the SF-36 questionnaire. F statistic (1,56) = 0.132
Statistical Analysis 15: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.574, ANOVA — Main effect of the Group x Visit interaction for the Social role area of the SF-36 questionnaire. F statistic (1,56) = 0.319
Statistical Analysis 16: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.490, ANOVA — Main effect of the Group for the Emotional role area of the SF-36 questionnaire. F statistic (1,56) = 0.482
Statistical Analysis 17: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.032, ANOVA — Main effect of the Visit for the Emotional role area of the SF-36 questionnaire. F statistic (1,56) = 4.850
Statistical Analysis 18: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.145, ANOVA — Main effect of the Group x Visit interaction for the Emotional role area of the SF-36 questionnaire. F statistic (1,56) = 2.181
Statistical Analysis 19: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.467, ANOVA — Main effect of the Group for the Mental health area of the SF-36 questionnaire. F statistic (1,56) = 0.535
Statistical Analysis 20: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.100, ANOVA — Main effect of the Visit for the Mental health area of the SF-36 questionnaire. F statistic (1,56) = 2.795
Statistical Analysis 21: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.890, ANOVA — Main effect of the Group x Visit interaction for the Mental health area of the SF-36 questionnaire. F statistic (1,56) = 0.019
Statistical Analysis 22: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.742, ANOVA — Main effect of the Group for the Physical Role area of the SF-36 questionnaire. F statistic (1,56) = 0.109
Statistical Analysis 23: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p < 0.001, ANOVA — Main effect of the Visit for the Physical Role area of the SF-36 questionnaire. F statistic (1,56) = 21.912. Effect size = 0.109
Statistical Analysis 24: Comparison: MBK-01 vs Fidaxomicin; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.089, ANOVA — Main effect of the Group x Visit interaction for the Physical Role area of the SF-36 questionnaire. F statistic (1,56) = 2.986

ADVERSE EVENTS:
Time Frame: Up to 6 months after the start of the treatment
Arm/Group | MBK-01 | Fidaxomicin
All-Cause Mortality (participants affected / at risk) | 1/45 | 1/47
Serious Adverse Events (participants affected / at risk) | 9/45 | 4/47
Other Adverse Events (participants affected / at risk) | 36/45 | 38/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBK-01 (N=45) | Fidaxomicin (N=47)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBK-01 (N=45) | Fidaxomicin (N=47)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dental discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 16 (17) | 22 (27)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (3)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Medical device site reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (3) | 1 (1)
Polyp (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 11 (13) | 6 (7)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 2 (2)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The statistical power of the study was limited due to the small sample size, which may have prevented finding statistically significant differences between MBK-01 and fidaxomicin.

Additionally, the lack of available comparative studies between FMT and fidaxomicin in primary episodes of CDI in the literature limits the ability to contextualize our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the results are not submitted by the sponsor, the PI may publish them in scientific journals, provided that they mention the sponsor, at least, within the first year after the authorization and marketing in any country (for non-commercialized products). The sponsor must receive for review a copy of the text, except otherwise agreed, at least 45 days before the submission (20 days before for Abstracts). The PI may only use these data with prior express written authorization from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT05201079/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT05201079/SAP_001.pdf